CLINICAL TRIAL: NCT05025345
Title: Clinical Evaluation of the Vision Performance of TECNIS EYHANCE™ Intraocular Lenses With TECNIS SIMPLICITY™ as Compared to TECNIS® 1-piece Intraocular Lenses
Brief Title: Vision Performance Evaluation of TECNIS EYHANCE™ With TECNIS SIMPLICITY™ Compared to TECNIS® 1-piece Intraocular Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMON-101-EHCE
Record Dates: First submitted 2021-08-26; First posted 2021-08-27 (Actual); Results first posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Study Lens (Experimental): Tecnis Eyhance
  Interventions: Device: Tecnis Eyhance
- Control Lens (Active Comparator): Tecnis 1 piece IOL (Intraocular lens)
  Interventions: Device: Tecnis 1 piece IOL

INTERVENTIONS:
Device: Tecnis Eyhance — Investigational intraocular lens replaces the natural lens removed during cataract surgery in both eyes.
  Arms: Study Lens
Device: Tecnis 1 piece IOL — Control intraocular lens replaces the natural lens removed during cataract surgery in both eyes.
  Arms: Control Lens

SUMMARY:
This study is a 6-month, prospective, multicenter, bilateral, randomized subject- and evaluator-masked, clinical investigation of the TECNIS Eyhance IOL versus the TECNIS 1-piece IOL.

The study will be conducted at up to 15 sites in the U.S.A and will enroll approximately 220 subjects to achieve approximately 200 randomized and bilaterally implanted subjects, resulting in approximately 100 evaluable subjects in each lens group at 6 months. Subjects are to be implanted with the same IOL in both eyes: TECNIS Eyhance IOL or the TECNIS 1-Piece IOL. The eye implanted first will be considered the primary study eye.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 22 years of age
* Bilateral cataracts for which posterior chamber IOL implantation has been planned
* Preoperative best corrected distance visual acuity (BCDVA) of 20/40 Snellen or worse with or without a glare source
* Potential for postoperative best corrected visual acuity of 20/30 Snellen or better
* Corneal astigmatism parameters:

  * Normal corneal topography and no irregular corneal astigmatism
  * Postoperative astigmatism can be surgically managed to be less than 1 D in each eye
* Clear intraocular media other than cataract in each eye
* Availability, willingness, ability, and sufficient cognitive awareness to comply with examination procedures and study visits
* Signed informed consent and HIPAA authorization or equivalent documentation necessary to comply with applicable privacy laws pertaining to medical treatment in the governing countries
* Ability to understand and respond to a questionnaire in English

Exclusion Criteria:

* Any conditions or circumstances, including those specified in the TECNIS Eyhance™ IOL Directions for Use, that, in the opinion of the investigator, may increase risk over benefit or result in an adverse event during the study.
* Inability to focus or fixate for prolonged periods of time (e.g., due to strabismus, nystagmus, etc.)
* Concurrent participation or participation within 60 days prior to preoperative visit in any other clinical trial
* Desire for monovision correction

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision Clinical Trials, Study Director — Johnson & Johnson Surgical Vision
Locations (15):
- United States (15):
  - Empire Eye & Laser Center, Bakersfield, California
  - Southern California Eye Physicians and Associates, Long Beach, California
  - Center For Sight, Sarasota, Florida
  - Jones Eye Clinic, Sioux City, Iowa
  - Chesapeake Eye Care & Laser Center, Annapolis, Maryland
  - Tekwani Vision Center, St Louis, Missouri
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - Eye Care Specialists, Kingston, Pennsylvania
  - Key-Whitman Eye Center, Dallas, Texas
  - Berkeley Eye Institute, P.A., Houston, Texas
  - Whitsett Vision Group, Houston, Texas
  - Texas Eye and Laser Center, Hurst, Texas
  - Focal Point Vision, San Antonio, Texas
  - Parkhurst NuVision, San Antonio, Texas
  - R & R Eye Research, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Devices Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 228 subjects were enrolled and 214 subjects were treated. Of the 214 subjects, 107 were implanted with the test lens and 107 with the control lens. 4 subjects did not complete the study.
Groups:
- Test Lens: Eyhance IOL, Model DIB00
- Control Lens: Monofocal IOL, Model ZCB00
Period: Overall Study
Arm/Group | Test Lens | Control Lens
Started | 107 | 107
Completed | 103 | 107
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Lens | Control Lens | Total
Number analyzed (Participants) | 107 | 107 | 214
Age, Customized [Number; unit: Participants]
  <60 | 9 | 8 | 17
  60-69 | 47 | 39 | 86
  70-79 | 42 | 51 | 93
  >=80 | 9 | 9 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 68 | 134
  Male | 41 | 39 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 15 | 33
  Not Hispanic or Latino | 89 | 92 | 181
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian (including Indian) | 4 | 1 | 5
  Black | 8 | 8 | 16
  Native Hawaiian/ Pacific Islander | 0 | 0 | 0
  Caucasian | 95 | 98 | 193
  Other Race | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: MONOCULAR BEST-CORRECTED DISTANCE VISUAL ACUITY (BCDVA)
Description: the mean monocular difference in Best-Corrected Distance Visual Acuity for the first eye between lens groups
Time Frame: 6 months
Population: The ITT (Intent-to-Treat) population for Monocular Best Corrected Distance Visual Acuity include all first eyes implanted with either a test or control IOL with data available at 6 months postoperative (i.e., no data imputation)
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: Eyes
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 103 | 107
Number analyzed (Eyes) | 103 | 107
LogMAR | -0.017 (0.090) | -0.029 (0.116)
Statistical Analysis 1: Comparison: Test Lens vs Control Lens; Test type: Non-Inferiority — Noninferiority margin equals -0.1; Success criteria was evaluated using lower confidence interval. No P-Value was calculated; Mean Difference (Final Values) = -0.013, 90% CI 2-sided [-0.036 to 0.011]

2. Secondary Outcome: MONOCULAR DISTANCE-CORRECTED INTERMEDIATE VISUAL ACUITY AT 66 CM (DCVA66)
Description: the mean monocular difference in Distance-Corrected Intermediate Visual Acuity at 66cm for first eyes between lens groups
Time Frame: 6 months
Population: The ITT (Intent-to-Treat) population for monocular first-eye distance-corrected intermediate visual acuity at 66cm (DCVA66) include all first eyes implanted with either a test or control IOL with data available at 6 months postoperative (i.e., no data imputation).
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: Eyes
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 103 | 107
Number analyzed (Eyes) | 103 | 107
LogMAR | 0.235 (0.169) | 0.348 (0.158)
Statistical Analysis 1: Comparison: Test Lens vs Control Lens; Test type: Superiority; p < 0.0001, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: During the course of the study until completion, 6 months.
Description: All adverse events (AEs), ocular and non-ocular, were monitored/assessed and planned to be reported for the first eye only. Second eye was not assessed for adverse events.
Arm/Group | Test Lens | Control Lens
All-Cause Mortality (participants affected / at risk) | 2/107 | 0/107
Serious Adverse Events (participants affected / at risk) | 5/107 | 4/107
Other Adverse Events (participants affected / at risk) | 1/107 | 0/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Lens (N=107) | Control Lens (N=107)
Cystoid macular edema (Eye disorders) | 1 (1) | 2 (4)
Lymphoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hospitalization (Surgical and medical procedures) | 1 (1) | 1 (1)
Refractory Cytopenia with Multilineage Dysplasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Mitral Valve Defect (Cardiac disorders) | 1 (1) | 0 (0)
Ischemic Optic Neuropathy (Eye disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Lens (N=107) | Control Lens (N=107)
Undesirable Optical Phenomena (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review results communication prior to public release and can embargo communications regarding trial results at anytime.

DOCUMENTS (2):
  • Study Protocol (2022-06-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT05025345/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT05025345/SAP_001.pdf